CLINICAL TRIAL: NCT00207987
Title: Changes in Cerebral Oxygenation During Deliberate Hypotensive Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Other Study IDs: DMR-93-41
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-11-21 (Estimated); Status verified 2005-09

CONDITIONS: Hypotension
Keywords: controlled hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This is a study using cerebral oximetry to evaluate the safety of traditionally adopted hypotensive anesthesia.

DETAILED DESCRIPTION:
The values of cerebral oximetry were analyzed between different stages of anesthetic management. The critical part of anesthetic management is to use the technique of controlled hypotension. The blood pressure was lowered to the level of MABP 50 or 60 mmHg depending on which group patients were assigned to.

The values of cerebral oximetry and side effects between 2 groups will be compared at the completion of data collection.

ELIGIBILITY:
Inclusion Criteria:

* 40 patients are going to receive complex spine surgery.

Exclusion Criteria:

* Neurologic diseases
* Hepatic or renal impairment
* Uncontrolled hypertension
* Cardiovascular diseases

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2003-10; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Yu C Liu, M.D., Principal Investigator — Anesthetic Department, China Medical University Hospital
Locations (1):
- Anesthetic Department, China Medical University Hospital, Taichung, Taiwan